CLINICAL TRIAL: NCT00217074
Title: Acupuncture for Hot Flashes: A Randomized Sham Controlled Clinical Study
Brief Title: Acupuncture and Hot Flashes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2294-03
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — Acupuncture Therapy

INTERVENTIONS:
Other: acupuncture

SUMMARY:
Methods: 103 participants, after being randomized to medical versus sham acupuncture received bi-weekly treatments for 5 weeks, after a baseline assessment week. They were then followed for an additional 7 weeks. Participants completed daily hot flash questionnaires, which formed the basis for analysis.

ELIGIBILITY:
Participants eligible for this study were females aged 45 to 59 with a reported average of ¡Ý 5 hot flashes a day

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2004-01; Primary Completion 2004-01 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Hot Flash Score

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States